CLINICAL TRIAL: NCT06027827
Title: Impact of Lateral Bone Grafting With Intraoperative Fusion in ACDF on Clinical Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XuanwuACDF
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: In addition to the central bone graft of the fusion cage, the lateral bone graft of the fusion cage was added.
  Interventions: Procedure: Addition of fusion device lateral bone graft
- control group: Conventional bone grafting in the center of the fusion

INTERVENTIONS:
Procedure: Addition of fusion device lateral bone graft — In addition to the central bone graft of the fusion cage, the lateral bone graft of the fusion cage was added.
  Groups: experimental group

SUMMARY:
The purpose of this trial was to investigate the safety and efficacy of fuser lateral bone grafting in ACDF. By observing the intervertebral bony fusion rate and clinical outcome scores of patients after fusion device lateral bone grafting, it was verified whether the fusion device lateral bone grafting approach could improve the bony fusion rate and clinical outcome of ACDF.

DETAILED DESCRIPTION:
The study will include patients who underwent 1-2 segment ACDF surgery, in addition to conventional surgical operations, the appropriate amount of allograft bone was implanted in the joint space of the hook vertebrae lateral to the fusion device, and X-rays and CTs were reviewed in the immediate postoperative period, March, June, and December, to verify intervertebral osseous fusion, as well as to observe the patient's clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years old; patients with cervical spondylosis who were about to undergo 1-2 segment ACDF surgery; agreement with the surgical plan and willingness to undergo long-term clinical follow-up; and signing of an informed consent form.

Exclusion Criteria:

* Drug or alcohol abusers; those with abnormal liver or kidney function unsuitable for surgery; those with cardiac insufficiency unsuitable for surgery; those with severe metabolic and endocrine diseases unsuitable for surgery; those with severe lung disorders such as asthma and abnormal lung function unsuitable for surgery; pregnant and breastfeeding women as well as those who are planning to become pregnant in the near future; those who have participated in other clinical trials within 3 months; and those who are not suitable for participation in the experiment in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Between the ages of 18-60 years; patients with cervical spondylosis about to undergo 1-2 segment ACDF surgery
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intervertebral bone fusion rate | 3rd month (±15 days), 6th month (±15 days), 1 year (±30 days) postoperatively
  primary Indicator

SECONDARY OUTCOMES:
JOA | Preoperative, 7 days postoperative, 3rd month (±15 days), 6th month (±15 days), 1 year (±30 days)
  Japanese Orthopaedic Association Scores

CONTACTS AND LOCATIONS:
Overall Officials: Fengzeng Jian, MD, PhD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Epstein NE. A Review of Complication Rates for Anterior Cervical Diskectomy and Fusion (ACDF). Surg Neurol Int. 2019 Jun 7;10:100. doi: 10.25259/SNI-191-2019. eCollection 2019. PMID 31528438
- [Result] Fountas KN, Kapsalaki EZ, Nikolakakos LG, Smisson HF, Johnston KW, Grigorian AA, Lee GP, Robinson JS Jr. Anterior cervical discectomy and fusion associated complications. Spine (Phila Pa 1976). 2007 Oct 1;32(21):2310-7. doi: 10.1097/BRS.0b013e318154c57e. PMID 17906571
- [Result] Wewel JT, Kasliwal MK, Adogwa O, Deutsch H, O'Toole JE, Traynelis VC. Fusion rate following three- and four-level ACDF using allograft and segmental instrumentation: A radiographic study. J Clin Neurosci. 2019 Apr;62:142-146. doi: 10.1016/j.jocn.2018.11.040. Epub 2019 Jan 25. PMID 30692036
- [Result] Godlewski B, Bebenek A, Dominiak M, Karpinski G, Cieslik P, Pawelczyk T. PEEK versus titanium-coated PEEK cervical cages: fusion rate. Acta Neurochir (Wien). 2022 Jun;164(6):1501-1507. doi: 10.1007/s00701-022-05217-7. Epub 2022 Apr 26. PMID 35471708
- [Result] Samartzis D, Shen FH, Lyon C, Phillips M, Goldberg EJ, An HS. Does rigid instrumentation increase the fusion rate in one-level anterior cervical discectomy and fusion? Spine J. 2004 Nov-Dec;4(6):636-43. doi: 10.1016/j.spinee.2004.04.010. PMID 15541695